CLINICAL TRIAL: NCT04520841
Title: Monocentric Randomized Clinical Trial Comparing Negative Pressure Wound Therapy (PREVENA™) and Standard Dry Dressings on Oozing of Closed Incision After Revision Total Hip and Knee Arthroplasty Surgery or Lower Extremity Amputation Surgery
Brief Title: Clinical Trial Comparing Negative Pressure Wound Therapy and Standard Dry Dressings
Acronym: BERLYTZ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Sylvain Steinmetz, Principal Investigator, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-00321
Record Dates: First submitted 2020-07-15; First posted 2020-08-20 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Arthroplasty Complications; Amputation; Prosthesis-Related Infections
Keywords: Prevena; Negative Pressure Wound Therapy; Revision Arthroplasty; Lower Extremity Amputation Surgery
MeSH Terms: conditions — Prosthesis-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard dry dressing in total hip or knee arthroplasty (Active Comparator): Standard dressing in total hip or knee arthroplasty surgery revision: a dry sterile dressing is applied on the surgical wound at the end of surgery
  Interventions: Device: Dry dressing
- Prevena in total hip or knee arthroplasty (Experimental): Prevena incision management system in total hip or knee arthroplastsy surgery revision:
  The Prevena incision management system is applied on the surgical wound at the end of surgery
  Interventions: Device: Prevena TM
- Standard dry dressing in lower limb amputation (Active Comparator): Standard dressing in lower limb amputation: a dry sterile dressing is applied on the surgical wound at the end of surgery
  Interventions: Device: Dry dressing
- Prevena in lower limb amputation (Experimental): Prevena incision management system in lower limb amputation:
  The Prevena incision management system is applied on the surgical wound at the end of surgery
  Interventions: Device: Prevena TM

INTERVENTIONS:
Device: Prevena TM — A Prevena Plus DuoTM Dressing Kit (KCI) is applied on the surgical wound at the end of surgery.
  Arms: Prevena in lower limb amputation; Prevena in total hip or knee arthroplasty
Device: Dry dressing — A standard dry sterile dressingwith non-adherent absorbent pad is applied on the surgical wound at the end of surgery
  Arms: Standard dry dressing in lower limb amputation; Standard dry dressing in total hip or knee arthroplasty

SUMMARY:
Negative pressure dressings are currently widely used in wound management. Their use is gradually being extended to surgical scars. However, studies demonstrating a clear benefit are rare, particularly in terms of postoperative discharge, the need for surgical revision due to prolonged oozing and cost.

The aim of this study is to evaluate the benefit of such a device in post-operative revision prosthesis surgery (hip and knee), as well as lower limb amputations.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years old
* Planned Surgery :

  1. revision of a hip or knee prosthesis, in 1 or 2 stages, at explantation and/or reimplantation, where
  2. elective amputation of a lower limb (transmetatarsal, trans-tibial (Burgess) or trans-femoral (Gritti-Stokes) level (nb: patients for whom amputation of both lower limbs is planned will be excluded)

Exclusion Criteria:

* Known allergy to dry dressings
* Patient already included in another clinical trial
* Inability to discern and/or inability to follow study procedures
* Known allergy to silver or another component of the system Prevena™
* Amputation for tumor pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Discharge after 7 days | Day 7- Day 8
  Presence of discharge at 7 days postoperatively (Day 7) Condition of the dry dressing applied on Day 7 and evaluated at least 24 hours after application (Day 8)

SECONDARY OUTCOMES:
Complications | Day 0 - Day 14
  Occurrence of post-operative complications from Day 0 to hospital discharge (or max Day 14)
Revision surgery | Day 0 - Day 14
  Occurrence of revision surgery due to persistent discharge from the day of the operation (Day 0) until discharge from hospital (or max Day 14)
Hospitalisation | Day 0 - Day 14
  Duration of hospitalisation from Day 0 to end of hospitalisation (in days)
Patient satisfaction | Day 7
  Reported patient satisfaction based on the responses obtained from the "Patient Evaluation Form" questionnaire completed by the patient. A numeric pain scale is included: the patient rates his pain on a scale of 0 to 10 when the last dry dressing (Opsite TM) is changed or when Prevena system (TM) is removed. Zero means "no pain," and 10 means "the worst possible pain."Participant will complete the questionnaire on Day 7.
Costs | Day 0 - Day 7
  Dressing repair costs (sum of the price of all dressings and materials needed for dressing repair) from Day 0 to Day 7 (in Swiss francs)
AE & ADE | Day 0 - Day 14
  Occurrence, intensity, severity, causal link with the medical device and the procedure, and characteristics of the adverse events (AEs) considered to be at least possibly related to the medical device or the procedure (= adverse events, ADEs), occurring from the day of the operation (Day 0) until discharge from hospital (or max Day 14).

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Steinmetz, MD, Principal Investigator — Lausanne University Hospital (Switzerland)
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided